CLINICAL TRIAL: NCT05299567
Title: Double-blind Placebo Trial to Determine the Efficacy and Safety of Treatment With Azithromycin for 6 Months in Patients With Post-infectious Bronchiolitis Obliterans
Brief Title: Efficacy and Safety of Azithromycin in Patients With Bronchiolitis Obliterans
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Claudio Castanos (Other Government)
Responsible Party: Sponsor-Investigator, Claudio Castanos, Head of Pediatric pulmonology, Hospital JP Garrahan
Organization: Hospital JP Garrahan (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 250463
Record Dates: First submitted 2017-05-18; First posted 2022-03-29 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-01

CONDITIONS: Bronchiolitis Obliterans
Keywords: bronchiolitis obliterans; Azithromycin
MeSH Terms: conditions — Bronchiolitis Obliterans | interventions — Azithromycin

STUDY DESIGN:
Intervention Model Description: Placebo-controlled, double-blind, randomized study
Who Masked: Care Provider, Investigator
Masking Description: Patients were randomly assigned by pharmacy staff in blocks of 4
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- azitrhomycin (Active Comparator): Group1 Azitrhomycin 250 or 500 mg in capsuls tree days a week for 6 months if the patiens are less or more than 40 kg respectively Exposure
  Interventions: Drug: Azithromycin
- Placebo (Placebo Comparator): Group 2 placebo Not exposure Placebo in capsuls tree days a week for 6 months
  Interventions: Drug: Azithromycin

INTERVENTIONS:
Drug: Azithromycin — Placebo with the same color and size than azithromycin tree days a wek for 6 months
  Other Names: placebo

SUMMARY:
Placebo-controlled, double-blind, randomized study. Post-infectious bronchiolitis obliterans (PIBO) patients aged 5 years and older of both sexes were enrolled.

DETAILED DESCRIPTION:
Bronchiolitis obliterans (BO) was defined as the presence of signs and symptoms of chronic obstructive lung disease: A) previously documented acute lower respiratory infection (ALRI) with persistence of airway obstruction and respiratory signs and symptoms, such as: dyspnea, tachypnea, retractions, persistent cough, increased antero-posterior diameter of the chest, persistent wheezing, crackles, exercise intolerance; B) findings such as: hyperinflation, atelectasis, and mosaic oligohemia on CT scan; and C) persistent obstructive pattern on pulmonary function test.

Patients were randomly assigned by pharmacy staff in blocks of 4 to receive either capsules of azithromycin 250 mg (Group 1) or placebo (Group 2) 3 days a week for 6 months. Patients whose weight was less than 40 kg received 250 mg 3 days a week (Monday, Wednesday, and Friday) and those weighing more than 40 kg received 500 mg in the same scheme, according to randomization to active drug or placebo. Pulmonary function and number of exacerbations were evaluated. Spirometry and plethysmography were performed at baseline and at 6 months. Variables analyzed were Forced vital capacity (FVC),Flow expiratory volume at the first second (FEV1), Total lung capacity (TLC),Residual volumen(RV),especific conductance (sGaw). Patients had been clinically stable over the previous three weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosis of Bronchiolitis obliternas
* older than 5 years
* Ability to perform pulmonary function test

Exclusion Criteria:

* Not being able to perform lung function study adequately
* Other causes of chronic lung disease (bronchopulmonary dysplasia, cystic fibrosis, primary or secondary immune deficiency)
* Previous history of portal hypertension, liver cirrhosis, splenomegaly or chang in normal values of laboratory at the start of the study.
* History of hypersensitivity to macrolides

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2010-08-24; Primary Completion 2011-07-21 (Actual); Study Completion 2011-07-21 (Actual)

PRIMARY OUTCOMES:
Percentages change in Forced Expiratory Volume in 1 second (FEV1) Number of Pulmonary exacerbation | 6 months
  1. FEV1 in percentages
  2. Pulmonary exacerbation in numbers

CONTACTS AND LOCATIONS:
Overall Officials: Claudio m Castaños, MD, Principal Investigator — Hospital de Pediatria "juan P. Garrahan"

IPD SHARING:
Plan to Share IPD: No